CLINICAL TRIAL: NCT03900546
Title: Influence of Arterial Tone Changes on Cardiac Output Measurement by Pressure Recording Analytical Method
Brief Title: Arterial Tone Influence on Cardiac Output Measured by PRAM
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Professor, Università Politecnica delle Marche
Other Study IDs: PRAM
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Output; Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MostCare — CO measurement using echocardiography and PRAM before and after noradrenaline dose change due to clinical reason

SUMMARY:
This study evaluates the role of arterial tone in the accuracy of cardiac output (CO) measurement by Pressure Recording Analytical Method (PRAM). Patients receiving noradrenaline who need for clinical reason to change the noradrenaline dose will be enrolled. We use echocardiography as reference method of CO measurement.

DETAILED DESCRIPTION:
Pressure Recording Analytical Method (PRAM) is an arterial pulse contour analysis method for CO measurement. As it is an uncalibrated method, one possible reason for its inaccuracy is rapid changes in arterial tone.

ELIGIBILITY:
Inclusion Criteria:

* invasive blood pressure monitoring on site
* need to start or change the dose of noradrenaline infusion for clinical reason

Exclusion Criteria:

* age <18
* arrhythmia
* severe valvular insufficiency
* pregnancy
* low quality arterial signal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to intensive care unit that need variation of noradrenaline dose for clinical reason.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Changes of cardiac output after variation of noradrenaline dose: ECO versus PRAM | Before and 30 minutes after noradrenaline dose variation
  Agreement between echocardiography and PRAM in CO measurement during arterial tone changes induced by different dose of noradrenaline

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, PhD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- Azienda Ospedaliero Universitaria Ospedali Riuniti Ancona, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.